CLINICAL TRIAL: NCT00379132
Title: A Phase I Imaging and Safety Study of Intravenous 131-I-TM-601 Labeled Chlorotoxin in Patients With Recurrent or Refractory Somatic and/or Cerebral Metastatic Solid Tumors
Brief Title: 131-I-TM-601 Study in Adults With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TransMolecular (Industry)
Responsible Party: Susan Stewart, Vice President, Regulatory Affairs, TransMolecular, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TM601-003
Record Dates: First submitted 2006-09-18; First posted 2006-09-21 (Estimated); Last update posted 2009-03-31 (Estimated); Status verified 2009-03

CONDITIONS: Breast Cancer; Non-Small Cell Lung Cancer; Melanoma; Colorectal Cancer; Pancreatic Cancer; Prostate Adenocarcinoma; Glioma; Primary Solid Tumors
Keywords: Glioma; prostatic; breast; non-small cell lung; melanoma; colorectal; pancreatic
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Melanoma; Colorectal Neoplasms; Pancreatic Neoplasms; Glioma | interventions — Chlorotoxin

INTERVENTIONS:
Drug: 131-I-TM-601 (chlorotoxin) — Patients will be administered 1 - 3 (Test Doses A, B, and Dose C) escalating doses of 131I-TM601 by intravenous (IV) administration. Each dose will be administered as a single administration, scheduled at one-week intervals.
  Test Dose A - 10 mCi (+/- 20%)/0.2 mg TM601 (131I-TM601) Test Dose B - 20 mCi (+/- 20%)/0.4 mg TM601 (131I-TM601) Dose C - 30 mCi (+/- 10%)/0.6 mg TM601 (131I-TM601)

SUMMARY:
This study is designed to evaluate the ability of intravenously (IV)administered 131-I-labeled TM-601 (chlorotoxin) to provide tumor-specific localization(via radiographic imaging) in patients with recurrent or refractory primary solid tumors with evidence of metastatic involvement. (Refractory tumors are non-responsive to standard treatment.) The safety and tolerability of IV administered 131-I-TM-601 in this patient population will be evaluated as part of this study.

DETAILED DESCRIPTION:
This is a multi-center, open label, non-randomized, sequential, within-patient dose-escalation study in patients with recurrent or refractory primary solid tumors with metastatic involvement (including brain metastases). Patients will be administered 1 to 3 (Test Doses A, B and Dose C) escalating doses of 131-I-TM-601 by intravenous (IV) administration, with dosimetry (imaging-based evaluation of the dose reaching the target sites) conducted prior to and following administration of each dose. Whole body dosimetry on critical structures including, but not limited to, bone marrow, bladder, brain, liver, and thyroid will be determined. The preliminary results from Test Dose Levels (A and/or B) for each patient will be analyzed prior to treating patients with Dose C.

Patients will be followed until 28 days following the final dose, with a complete clinical assessment and imaging evaluations at the final follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed recurrent or refractory primary solid tumor malignancy. Primary tumor cell type is one of the following: breast, non-small cell lung, melanoma, colorectal, prostatic adenocarcinoma (hormone refractory) or glioma. Note: Patients with a primary solid tumor cell type not listed above, meeting all other selection criteria may be considered eligible, on a case by case basis
* Demonstration of distant metastatic involvement as seen with standard clinical non-invasive imaging techniques (CT/MRI) or on biopsy. Note: on a case-by-case basis, patients with a locally recurrent, unresectable (inoperable) tumor may be considered for inclusion
* Refractory to standard curative treatment
* At least 18 years of age
* Baseline Karnofsky Performance Status (KPS) of 60-100%
* Life expectancy, based on investigator judgement, of greater than 3 months
* Adequate organ and marrow function (as defined in protocol)
* Women of child-bearing potential must have a negative pregnancy test, refrain from nursing, and must agree to use appropriate contraception for the duration of the trial

Exclusion Criteria:

* Prior cytotoxic chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Patients who have not sufficiently recovered from adverse events due to previously administered agents
* Concurrent treatment with investigational or commercial agents or therapies administered with the intent to treat the patient's malignancy, including chemotherapy, immunotherapy, biological response modifiers, or palliative radiotherapy. Possible exceptions (at the discretion of the investigator) are for hormonal therapy for breast and prostate cancer, hematologic, analgesic, biphosphonate, and any other form of supportive therapy.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 131-I-labeled chlorotoxin (e.g. iodine or iodine-containing drugs)
* Patients with uncontrolled intercurrent illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-08; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To evaluate whether intravenous (IV) 131-I-TM-601 provides tumor-specific localization in patients with recurrent or refractory metastatic (including brain metastases) solid tumors | between 1 - 72 hours post study dose
To determine the distribution and dosimetry of intravenously administered 131-I-TM-601 | between 1 - 72 hours post study dose
To determine the safety and tolerability of IV administered 131-I-TM-601. | within 28 days of last study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: John Fiveash, MD, Principal Investigator — University of Alabama at Birmingham; Jeffrey Raizer, M.D., Principal Investigator — Northwestern University; Neil Senzer, MD, Principal Investigator — Mary Crowley Medical Research Center; Thomas Gribbins, MD, Principal Investigator — Lacks Cancer Center at St. Mary's Health Care; Jay-Jiguang Zhu, MD, Principal Investigator — Tufts Medical Center; Steven Chmura, MD, Principal Investigator — University of Chicago
Locations (6):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Northwestern University, The Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Tufts - New England Medical Center, Boston, Massachusetts
  - Lacks Cancer Center at St. Mary's Health Care, Grand Rapids, Michigan
  - Mary Crowley Medical Research Center, Dallas, Texas

REFERENCES:
- [Background] Mamelak AN, Jacoby DB. Targeted delivery of antitumoral therapy to glioma and other malignancies with synthetic chlorotoxin (TM-601). Expert Opin Drug Deliv. 2007 Mar;4(2):175-86. doi: 10.1517/17425247.4.2.175. PMID 17335414
- [Background] Mamelak AN, Rosenfeld S, Bucholz R, Raubitschek A, Nabors LB, Fiveash JB, Shen S, Khazaeli MB, Colcher D, Liu A, Osman M, Guthrie B, Schade-Bijur S, Hablitz DM, Alvarez VL, Gonda MA. Phase I single-dose study of intracavitary-administered iodine-131-TM-601 in adults with recurrent high-grade glioma. J Clin Oncol. 2006 Aug 1;24(22):3644-50. doi: 10.1200/JCO.2005.05.4569. PMID 16877732
- [Background] Hockaday DC, Shen S, Fiveash J, Raubitschek A, Colcher D, Liu A, Alvarez V, Mamelak AN. Imaging glioma extent with 131I-TM-601. J Nucl Med. 2005 Apr;46(4):580-6. PMID 15809479
- [Background] Lyons SA, O'Neal J, Sontheimer H. Chlorotoxin, a scorpion-derived peptide, specifically binds to gliomas and tumors of neuroectodermal origin. Glia. 2002 Aug;39(2):162-73. doi: 10.1002/glia.10083. PMID 12112367